CLINICAL TRIAL: NCT04011527
Title: A Prospective Follow-up Assessment in Bad Segeberg With Patients Undergoing a Rotational Atherectomy in Coronary Lesion/s
Brief Title: The Prospective Segeberg Registry for Rotational Atherectomy in Coronary Lesion/s
Status: Recruiting | Type: Observational
Sponsor: Segeberger Kliniken GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: SK 111 -- 168/11
Record Dates: First submitted 2019-06-28; First posted 2019-07-08 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease
Keywords: Calcified coronary artery lesions
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atherectomy, Coronary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Coronary Artery Disease: Patients with Coronary Artery Disease undergoing a Rotational Atherectomy in Coronary Lesion/s
  Interventions: Procedure: Rotational Atherectomy in Coronary Lesion/s

INTERVENTIONS:
Procedure: Rotational Atherectomy in Coronary Lesion/s

SUMMARY:
A Prospective Follow-up Assessment in Bad Segeberg with Patients undergoing a Rotational Atherectomy in Coronary Lesion/s

DETAILED DESCRIPTION:
A prospective single center registry including all patients treated with Rotational Atherectomy in Coronary Lesion/s at the Heart Center, Bad Segeberg, Germany. Patients undergo a routine clinical follow-up schedule, including a long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a rotational atherectomy of coronary lesion/s

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease undergoing a rotational atherectomy in coronary lesion/s
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2002-11-25 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of in-hospital and long-term cardiovascular adverse events in percent | 2 years
  Peri-procedural events and in-hospital cardiovascular events and long-term cardiovascular events (bleeding, peripheral and coronary vascular complication, stroke, myocardial infarction, stent thrombosis, revascularization, death)

CONTACTS AND LOCATIONS:
Overall Officials: Gert Richardt, Prof., MD, Study Director — Herzzentrum Segeberger Kliniken GmbH
Locations (1):
- Herzzentrum Segeberger Kliniken GmbH, Bad Segeberg, Germany